CLINICAL TRIAL: NCT07074002
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate the Efficacy and Safety of BP1.4979 in Adult Patients With Essential Tremor
Brief Title: Proof of Concept Study on BP1.4979 Effect on Essential Tremor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P23-05/BP1.4979
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Essential Tremor
Keywords: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: Multicentre, randomised, double-blind, placebo-controlled, parallel-group trial, proof of concept study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BP1.4979 (Experimental): One tablet of BP1.4979 taken twice daily for 4 weeks, approximately 8 to 10 hours apart
  Interventions: Drug: BP1.4979
- Placebo (Placebo Comparator): One tablet of placebo taken twice daily for 4 weeks, approximately 8 to 10 hours apart
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BP1.4979 — Selective dopamine D3 partial agonist
  Arms: BP1.4979
Drug: Placebo — Matching placebo of BP1.4979 tablet
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if drug BP1.4979 works to treat essential tremors in adults. It will also learn about the safety of drug BP1.4979. The main questions it aims to answer are:

* Does the drug BP1.4979 reduce tremors in individuals with essential tremor?
* Do participants have a good safety and tolerability of drug BP1.4979?

Researchers will compare drug BP1.4979 to a placebo (a look-alike substance that contains no drug) to see if drug BP1.4979 works to treat essential tremors.

Participants will:

* Take the study drug (active or a placebo) twice daily over a 4-week period
* Visit the clinic 5 times for health checkups and questionnaires completion over a period of approximately 7 to 10 weeks
* Complete a diary weekly to assess the impact of essential tremor on daily life

DETAILED DESCRIPTION:
Essential tremor (ET) is the most common form of movement-related tremor, affecting approximately 1% of the global population and up to 5% of individuals over 60 years old. This condition significantly impacts quality of life, as it often makes daily tasks difficult to perform.

Current treatments, mainly beta-blockers (e.g., propranolol), do not work for everyone and often cause bothersome side effects.

The exact causes of ET remain poorly understood, suggesting that it may be a syndrome (a group of related disorders) rather than a single disease. Brain imaging studies show that certain parts of the brain responsible for movement do not function normally, but it is not yet clear whether this is a disease that worsens over time.

Researchers believe that the brain chemical dopamine plays a key role in ET. One of dopamine receptors could be an interesting target for treatment. Drugs acting on this receptor have already shown positive results in other conditions, such as Parkinson's disease.

The objective of this trial is to develop a more effective treatment for ET, addressing an unmet medical need and improving the quality of life of affected patients.

The study drug, BP1.4979, acts on the dopamine pathway and is being tested to assess whether it can reduce tremors in individuals with ET. The study will compare BP1.4979 to a placebo (an identical-looking tablet with no active ingredient), taken twice daily over a 4-week period.

The study is a double-blind trial compared to a placebo, which means that neither the participants nor the study doctors know who is receiving the study drug or the placebo so as not to influence the results obtained. The treatments will be assigned randomly (by drawing lots), thus forming one group receiving BP1.4979 (20 mg) and another receiving the corresponding placebo.

A visit to the clinical site will take place at the beginning of the screening phase. Participants will be asked to sign an informed consent form before any study-related procedures.

Patients will then return to the clinical site to check whether they are eligible to take part in the study during the "randomization visit", and if so, they will receive study drug for 4 weeks of treatment.

Patients will be asked to complete a questionnaire once a week during the treatment period, to assess the impact of tremor on daily life.

Follow-up visits will take place every 2 weeks thereafter, at Week 2 (safety assessments) and Week 4 (end-of-treatment visit). A final visit will be made at Week 6 (15 days after stopping treatment) to check for or monitor any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18-85 years old
* Confirmed diagnosis of ET, characterized by meeting the following criteria: (a) the presence of a bilateral upper limb action tremor that occurs in isolation; (b) a minimum duration of 3 years; and (c) the tremor may or may not be present in other areas such as the voice, or lower limbs
* ET characterized by a TETRAS-P score of at least 1.5 in either the forward posture, wing beating posture, or finger-to-nose movement of at least one upper extremity
* Female patient: post-menopausal woman having at least 12 months of natural amenorrhea without any alternative medical cause, or woman of childbearing potential using a highly effective method of contraception for the duration of the trial and for 1 month after stopping the investigational medication

Exclusion Criteria:

* Severe tremor, defined as patient with ET characterized by a TETRAS-P score of ≥ 3 in either the forward posture, wing beating posture, or finger-to-nose movement of at least one upper extremity, or tremor of trunk
* Isolated head tremor not accompanied with tremor of any other body part
* Medical history or clinical evidence of any other conditions, whether medical, neurological, or psychiatric, that could potentially explain or contribute to the presence of tremors
* Patient who takes a medication which may induce tremor
* Direct or indirect injury or trauma to the nervous system within 3 months before the onset of tremor
* Concomitant treatment with more than three drugs to treat ET
* Any prior procedures for the treatment of ET such as deep brain stimulation, brain lesioning, or magnetic resonance (MR)-guided procedures, including MR-guided focused ultrasound

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Performance Subscale of The Essential Tremor Rating Assessment Scale (TETRAS-P) | 4 weeks
  Change in the total score of the Performance Subscale of The Essential Tremor Rating Assessment Scale (TETRAS-P) after 4 weeks of treatment.

OTHER OUTCOMES:
Global satisfaction questionnaire | 4 weeks
  Assessment of patient satisfaction with the study drug compared to any previously used anti-tremor medication via the global satisfaction questionnaire.
Patient reported outcome (PRO) | 4 weeks
  Change in patient's experience via the patient reported outcome (PRO) assessing the impact of essential tremors on daily living.

CONTACTS AND LOCATIONS:
Overall Officials: David Devos Coordinating Investigator, Pr, Principal Investigator — CHU de Lille
Locations (14):
- France (14):
  - CHU Amiens-Picardie, Amiens
  - CHU Besançon, Besançon
  - Hospices Civils De Lyon Hôpital Neurologique Pierre Wertheimer, Bron
  - CHU de Clermont-Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU Henri Mondor, Créteil
  - CHU de Lille - Hôpital Roger SALENGRO, Lille
  - Centre Hospitalier Régional De Marseille - Hôpital de la Timone, Marseille
  - CHRU Nancy - Hôpital Central, Nancy
  - CHU de Nice - Hôpital Pasteur 2, Nice
  - CHU de Nîmes, Nîmes
  - CHU Poitiers, Poitiers
  - CHU Rennes - CHU Pontchaillou, Rennes
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHU Purpan - Bâtiment Pierre Paul Riquet, Toulouse

IPD SHARING:
Plan to Share IPD: No